CLINICAL TRIAL: NCT00971620
Title: Randomized Pilot Study for the Treatment of Cutaneous Leiomyomas With Botulinum Toxin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edward Cowen, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 090072; 09-C-0072; NCT00842725 (obsolete NCT alias)
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Cutaneous Leiomyomas; Hereditary Leiomyomatosis and Renal Cell Cancer
Keywords: Cutaneous Leiomyomas; Skin Pain; Botox Therapy; Hereditary Leiomyomatosis; Renal Cell Cancer; Cutaneous Leiomyoma
MeSH Terms: conditions — Hereditary leiomyomatosis and renal cell cancer; Carcinoma, Renal Cell | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BTX-A (Experimental): BTX-A intralesional injection
  Interventions: Biological: Botulinum toxin type A
- Placebo/Saline (Experimental): Saline intralesional injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — Given as an intralesional injection.
  Other Names: BTX-A
  Arms: BTX-A
Other: Placebo — Given as an intralesional injection
  Arms: Placebo/Saline

SUMMARY:
Cutaneous leiomyomas are benign tumors of smooth muscle origin. They can be very painful, and current treatments for the tumors and for the associated pain do not produce satisfactory results. One potential treatment for localized severe muscle pain involves injections with botulinum toxin A. This study will investigate the effectiveness, side effects, and dosage of botulinum toxin A (BOTOX) as a treatment for patients with pain associated with cutaneous leiomyomas.

This study will include 18 subjects, all of whom will be 18 years of age and older, who have pain associated with cutaneous leiomyomas.

For the 24-week study, patients will be randomly assigned to one of two treatment groups. Neither the study team nor the patient will know to which group patients have been assigned. Before the study begins, all participants must provide a full medical history for research and evaluation purposes, fill out pain and quality-of-life questionnaires, and undergo an ice test in which researchers will apply ice to the site of the cutaneous leiomyomas and ask participants to evaluate the level of pain before and after ice application. Both groups will be required to keep a pain diary throughout the study to record their level of pain on a daily basis, and will be asked to avoid or restrict the use of specific medications or other remedies to treat the pain.

At the first visit (Week 0), one group will receive a prescribed dose of botulinum toxin A, which will be administered as an injection into the leiomyoma, and the other (control) group will receive a placebo injection of a saline solution. Patients will return 4 weeks later, at which time they will undergo a medical examination, and the ice test, and complete questionnaires to assess responses and level of pain. Patients will return in Week 12, at which time the group assignment will be revealed (un-blinded) to investigators and patients. Patients who received placebo injections will be offered the opportunity to receive injection of botulinum toxin A into their leiomyomas. All patients will undergo a medical examination, the ice test, complete questionnaires, and continue completing their daily pain diaries at home. The final visit, in Week 24, will follow the same procedure as the Week 4 visit.

At the end of the study, patients may be eligible to have one or more of the painful cutaneous leiomyomas surgically removed if the researchers believe that the skin lesions can be removed with a reasonable cosmetic result.

DETAILED DESCRIPTION:
Background:

* Cutaneous leiomyomas are smooth muscle tumors that may arise sporadically or in association with an inherited cancer-related genodermatosis.
* Leiomyomas may be severely painful, and current management is generally unsatisfactory.
* Studies demonstrate increased nerve density within and around leiomyomas as well as increased acetylcholinesterase staining of associated nerves.
* Botulinum toxin-A has been used in the treatment of pain syndromes.
* Based on the known mechanisms of action of botulinum toxin-A, treatment with botulinum toxin-A (BOTOX; Allergan, Inc.), may ameliorate the severe paroxysmal pain of symptomatic cutaneous leiomyomas.

Objectives:

* Primary: To assess change in worst lesional pain in the past week based on Brief Pain Inventory (BPI) from Week 0 to Week 4 in treated patients versus controls.
* Primary: To assess improvement in pain based on Visual Analog Scale (VAS) after application of ice at Week 4 compared to baseline in treated patients versus controls.
* Secondary: To assess change in magnitude and in frequency of painful episodes based on a weekly patient diary in treated patients versus controls.
* Secondary: To assess persistence of pain control at Weeks 12 based on the BPI and VAS.
* Secondary: To assess the frequency of rescue pain medication use in treated patients versus controls during the 24 week study period.
* Secondary: To determine the impact of leiomyoma treatment on quality of life.
* Secondary: To assess change in patient s condition based on the Patient Global Impression of Change.
* Secondary: To evaluate the immunohistochemical staining of nerve fibers and muscle in cutaneous leiomyomas in control and treated lesions following the conclusion of the study.

Eligibility:

* Subjects greater than or equal to18 years with at least 1 symptomatic cutaneous leiomyoma.
* Pain symptoms must occur at least once a week and be characterized as greater than or equal to 5 out of 10.

Design:

* A 12-week double-blind placebo controlled pilot study of 18 subjects with symptomatic leiomyomas will include initial assessment with BPI, photography, and skin biopsies, followed by treatment of subjects who initially received placebo.
* Cutaneous leiomyomas will undergo intralesional injection with botulinum toxin-A.
* Subjects will return at Weeks 4 and 12 for repeat assessment using pain and quality of life questionnaires and photography. Skin biopsies will be performed at week 12.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Subjects must be age greater than or equal to18 years.
  2. Subjects must have a prior biopsy-proven diagnosis of cutaneous leiomyoma.
  3. Subjects must have at least 1 symptomatic leiomyomas or regions less than or equal to 60 cm^2 of leiomyomas with pain characterized as greater than 4 based on a 10-point scale, indicating pain of at least moderate severity.
  4. Pain episodes must occur at least once a week.
  5. Subjects must have the ability to participate fully and comply with the procedures of the protocol in the opinion of the investigator.
  6. Written informed consent has been obtained including consenting to have tissue samples stored, however subjects are allowed to refuse sample storage.
  7. Negative urine or serum pregnancy test in females of childbearing potential.
  8. Subjects who are clinically stable such that they can be expected to complete the 24-week study.

EXCLUSION CRITERIA:

1. Subjects with allergies to BTX-A.
2. Females with a positive pregnancy test, or who are breast-feeding, planning a pregnancy during the study, who think that they may be pregnant at the start of the study or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study.
3. Subjects with neuromuscular junction disorders (ie. myasthenia gravis or Lambert-Eaton syndrome) or peripheral motor neuropathic diseases (ie. amyotrophic lateral sclerosis or motor neuropathy).
4. Subjects with infection at the intended sites of injection.
5. Subjects who have had prior Botulinum toxin product within the past 6 months.
6. Subjects with pain resulting from other disease(s), specifically:

   * pain that requires intermittent or ongoing treatment with narcotics
   * severe, debilitating, or acute pain originating from sources other than leiomyomas
7. Subjects taking pain medications, neuroactive agents, or other therapy directed toward treatment of cutaneous leiomyomas concurrently or within 5 days or 5 half-lives (whichever is longer) of BTX-A treatment, other than specified rescue pain medications). Patients currently on therapy directed toward OTHER mild to moderate chronic pain will be evaluated on a case-by-case basis for inclusion. Patients with well-controlled mild to moderate chronic pain such as that associated with osteoarthritis, who do not require narcotic therapy, will NOT be excluded. Aspirin for pain relief or for other indications is also acceptable.
8. Subjects with late-stage cancers or unstable disease (such as hemodynamic instability, i.e., systolic or diastolic blood pressure fall of 20 mm Hg or greater from the stable patient s baseline measurement).
9. A condition or situation that, in the investigator's opinion, may put the subject at significant risk or interfere significantly with the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-11-17 (Actual); Primary Completion 2014-01-09 (Actual); Study Completion 2016-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward W Cowen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Archer CB, Whittaker S, Greaves MW. Pharmacological modulation of cold-induced pain in cutaneous leiomyomata. Br J Dermatol. 1988 Feb;118(2):255-60. doi: 10.1111/j.1365-2133.1988.tb01783.x. PMID 3348971
- [Background] Batchelor RJ, Lyon CC, Highet AS. Successful treatment of pain in two patients with cutaneous leiomyomata with the oral alpha-1 adrenoceptor antagonist, doxazosin. Br J Dermatol. 2004 Apr;150(4):775-6. doi: 10.1111/j.0007-0963.2004.05880.x. No abstract available. PMID 15099382
- [Background] Raj S, Calonje E, Kraus M, Kavanagh G, Newman PL, Fletcher CD. Cutaneous pilar leiomyoma: clinicopathologic analysis of 53 lesions in 45 patients. Am J Dermatopathol. 1997 Feb;19(1):2-9. doi: 10.1097/00000372-199702000-00002. PMID 9056647
- [Result] Naik HB, Steinberg SM, Middelton LA, Hewitt SM, Zuo RC, Linehan WM, Kong HH, Cowen EW. Efficacy of Intralesional Botulinum Toxin A for Treatment of Painful Cutaneous Leiomyomas: A Randomized Clinical Trial. JAMA Dermatol. 2015 Oct;151(10):1096-102. doi: 10.1001/jamadermatol.2015.1793. PMID 26244563
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0072.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BTX-A | Placebo/Saline
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BTX-A | Placebo/Saline | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (15.6) | 45.5 (11.4) | 47.0 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18
Leiomyoma Distribution [Count of Participants; unit: Participants]
  Single | 1 | 3 | 4
  Segmental | 7 | 6 | 13
  Disseminated | 1 | 0 | 1
Location of Lesions [Count of Participants; unit: Participants]
  Neck | 1 | 0 | 1
  Torso | 6 | 4 | 10
  Extremity | 2 | 5 | 7
Volume of Drug Administered [Mean (Standard Deviation); unit: mL] | 2.41 (0.70) | 1.12 (0.38) | 1.76 (.54)

OUTCOME MEASURES:

1. Primary Outcome: Change in Worst Lesional Pain in the Past Week Based on Brief Pain Inventory
Description: Change in worst lesional pain in the past week based on Brief Pain Inventory (BPI) from Week 0 to Week 4 in treated patients versus controls. The BPI uses an arbitrary units on a 0-10 scale. For the purposes of the statistical calculation, a difference of 1 standard deviation between groups at baseline vs. week 4 was considered significant. Any BPI value above zero (no pain) is abnormal. The mean change indicates mean change in pain score.
Time Frame: Between week 0 and week 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BTX-A | Placebo/Saline
Number analyzed (Participants) | 9 | 9
units on a scale | -2.50 (0.46) | -1.26 (0.53)

2. Primary Outcome: Median Change in Average Pain Between Two Arms
Description: Change in average pain was assessed by the Brief Pain Inventory (BPI). The BPI is a validated pain assessment tool that assesses severity of pain, location of pain, impact of pain on daily functions, pain medications, and amount of pain relief in the past 24 hours or past week (e.g. scale of 0-10 (worst pain)).
Time Frame: Between weeks 0 and week 4
Measure: Median (Full Range); unit: Score
Arm/Group | BTX-A | Placebo/Saline
Number analyzed (Participants) | 9 | 9
Score | 0.00 [-6.00 to 2.00] | 0.00 [-5.00 to 3.00]
Statistical Analysis 1: Comparison: BTX-A vs Placebo/Saline; Test type: Superiority or Other; p = .70, Wilcoxon rank sum test; Hodges-Lehmann = 0.00, 95% CI 2-sided [-2.00 to 4.00]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 37 months
Measure: Number; unit: participants
Arm/Group | BTX-A | Placebo/Saline
Number analyzed (Participants) | 9 | 9
participants | 4 | 5

4. Secondary Outcome: Visual Analog Scale (VAS) of Patient Perceived Pain at Leiomyoma Site Prior to Ice Provocation at Week 0 vs. Week 4
Description: The VAS is a commonly used validated tool for assessment of pain. For this measure, a 10-cm VAS was used to assess current patient pain/discomfort before application of ice to study lesions at week 0 and week 4. A clinically meaningful change in chronic pain intensity using the VAS has been determined as a reduction of 2 points or 30%. Range is 0-10; 0 is no pain and 10 is worst possible pain.
Time Frame: Week 0 vs. week 4
Measure: Median (Full Range); unit: Score
Arm/Group | BTX-A | Placebo/Saline
Number analyzed (Participants) | 9 | 9
Score | 0.00 [-3.30 to 0.70] | 0.40 [-1.30 to 1.50]
Statistical Analysis 1: Comparison: BTX-A vs Placebo/Saline; Test type: Superiority or Other; p = .06, Wilcoxon rank sum test

5. Secondary Outcome: Comparison of Change in Skin Related Quality of Life by Total Dermatology Life Quality Index (DLQI) at Week 0 vs. Week 4
Description: The DLQI is a 10-question quality of life survey which has been extensively validated and frequently used in dermatologic disorders such as atopic dermatitis, acne, and psoriasis. Score is 0-30 based on 10 questions. The higher the score, the more quality of life is impaired.
Time Frame: Week 0 vs. week 4
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | BTX-A | Placebo/Saline
Number analyzed (Participants) | 9 | 9
Units on a scale | -4.00 [-8.00 to 2.00] | 0.00 [-1.00 to 4.00]
Statistical Analysis 1: Comparison: BTX-A vs Placebo/Saline; Test type: Superiority or Other; p = .007, WIlcoxon rank sum test

6. Secondary Outcome: Specific Skin Pain-Related Question on the Dermatology Life Quality Index
Description: The DLQI is a 10-question quality of life survey which has been extensively validated and frequently used in dermatologic disorders such as atopic dermatitis, acne, and psoriasis. Participants response to the question "Over the last week, how itchy, sore, painful or stinging has your skin been?" was assessed by the Dermatology Life Quality Index. This outcome refers to a single specific question on the DLQI, so the range for this outcome is 0-3. Lower values in the DLQI indicate less impairment (or greater improvement) in life quality from the skin disease.
Time Frame: Week 0 vs. week 4
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | BTX-A | Placebo/Saline
Number analyzed (Participants) | 9 | 9
Units on a scale | -1.00 [-2.00 to 1.00] | 0.00 [-1.00 to 0.00]
Statistical Analysis 1: Comparison: BTX-A vs Placebo/Saline; Test type: Superiority or Other; p = 0.48, Wilcoxon rank sum test

7. Secondary Outcome: Change in Post-Ice Provocation Visual Analog Score (VAS) Between Week 12 and Week 24
Description: The VAS is a commonly used validated tool for assessment of pain. The 10-cm VAS was used to assess current patient pain/discomfort before and after application of ice to study lesions. A clinically meaningful change in chronic pain intensity using the VAS has been determined as a reduction of 2 points or 30%. Scale is 0-10. 10 denotes worse pain than 0.
Time Frame: Between week 12 and 24
Measure: Median (Full Range); unit: Score
Arm/Group | BTX-A | Placebo/Saline
Number analyzed (Participants) | 9 | 9
Score | 4.10 [2.50 to 5.90] | -0.30 [-8.50 to 1.10]
Statistical Analysis 1: Comparison: BTX-A vs Placebo/Saline; Test type: Superiority or Other; p = .04, Wilcoxon rank sum test

8. Secondary Outcome: Immunohistochemical Staining of Cutaneous Leiomyomas for Acetylcholinesterase (AchE) Before (i.e.,Week 0) and 12 Weeks After Botulinum Toxin Administration
Description: AchE staining was scored as 0 (none), 1 (rare), 2 (scattered), or 3 (focal or greater).
Time Frame: Week 0 vs. week 12
Measure: Median (Full Range); unit: Score
Arm/Group | BTX-A | Placebo/Saline
Number analyzed (Participants) | 9 | 9
Score | 1.00 [0.00 to 2.00] | 0.00 [-1.00 to 0.00]

9. Secondary Outcome: Immunohistochemical Staining of Cutaneous Leiomyomas for C-fos Before (i.e., Week 0) and 12 Weeks After Botulinum Toxin Administration
Description: c-fos, a marker of neuronal activation after pain stimulation, was scored as 0 (none), 1 (scattered), 2 (<66% of tumor cells), or 3 (≥66% of tumor cells).
Time Frame: Week 0 vs. week 12
Measure: Median (Full Range); unit: Score
Arm/Group | BTX-A | Placebo/Saline
Number analyzed (Participants) | 9 | 9
Score | -1.00 [-1.00 to 0.00] | 0.00 [0.00 to 1.00]
Statistical Analysis 1: Comparison: BTX-A vs Placebo/Saline; Test type: Superiority or Other; p = .07, Wilcoxon rank sum test

10. Secondary Outcome: Percentage of Patients With a Change in Average Pain Score
Description: Average pain was determined from a 0-10 scale question on the Brief Pain Inventory (BPI). 10 denotes worse pain.
Time Frame: Week 0 score vs. week 4 score
Measure: Number; unit: percentage of patients
Arm/Group | BTX-A | Placebo/Saline
Number analyzed (Participants) | 9 | 9
percentage of patients
  >50% pain reduction | 44 | 22
  ≤50% pain reduction | 0 | 11
  No change in pain | 22 | 33
  Increased pain | 22 | 22
  Missing | 11 | 11

11. Secondary Outcome: Percentage of Patients With a Change in Pre-Ice Visual Analog Score (VAS) Between Week 0 and Week 4
Description: The VAS is a commonly used validated tool for assessment of pain. The 10-cm VAS was used to assess current patient pain/discomfort before and after application of ice to study lesions. A clinically meaningful change in chronic pain intensity using the VAS has been determined as a reduction of 2 points or 30%. Scale of 0-10. 10 = worse pain.
Time Frame: Week 0 vs. week 4
Measure: Number; unit: percentage of patients
Arm/Group | BTX-A | Placebo/Saline
Number analyzed (Participants) | 9 | 9
percentage of patients
  >50% pain reduction | 22 | 11
  ≤50% pain reduction | 33 | 0
  No change in pain | 0 | 11
  Increased pain | 11 | 55
  Missing | 33 | 22

12. Secondary Outcome: Percentage of Patients With a Change in Post-Ice Visual Analog Score (VAS) Between Week 0 and Week 4
Description: The VAS is a commonly used validated tool for assessment of pain. The 10-cm VAS was used to assess current patient pain/discomfort before and after application of ice to study lesions. A clinically meaningful change in chronic pain intensity using the VAS has been determined as a reduction of 2 points or 30%. Scale is 0-10. 10 = worse pain.
Time Frame: Week 0 vs. week 4
Measure: Number; unit: percentage of patients
Arm/Group | BTX-A | Placebo/Saline
Number analyzed (Participants) | 9 | 9
percentage of patients
  >50% pain reduction | 33 | 33
  ≤50% pain reduction | 44 | 44
  No change in pain | 0 | 0
  Increased pain | 22 | 22
  Missing | 0 | 0

13. Secondary Outcome: Worst Pain Severity
Description: Pain severity was assessed by the Brief Pain Inventory (BPI). The BPI is a validated pain assessment tool that assesses severity of pain, location of pain, impact of pain on daily functions, pain medications, and amount of pain relief in the past 24 hours or past week (e.g. scale of 0-10 (worst pain)). This outcome was based on a single 0-10 question on the BPI.
Time Frame: Week 0 vs. week 4
Measure: Median (Full Range); unit: Score
Arm/Group | BTX-A | Placebo/Saline
Number analyzed (Participants) | 9 | 9
Score | -2.25 [-5.00 to 0.25] | -0.75 [-3.75 to 0.50]

ADVERSE EVENTS:
Time Frame: 37 months
Description: There are no unexpected adverse events at grade 2 or higher.
Arm/Group | BTX-A | Placebo/Saline
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 4/9 | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BTX-A (N=9) | Placebo/Saline (N=9)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 0 (0) | 1 (1)
Constitutional Symptoms - Other (Specify, __) (General disorders) | 1 (1) | 1 (1) — BTX-A: Sinus congestion; Placebo: Sore throat
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bronchus (Infections and infestations) | 1 (1) | 0
Infection with normal ANC or Grade 1 or 2 neutrophils::Sinus (Infections and infestations) | 0 | 1 (1)
Infection with unknown ANC::Upper airway NOS (Infections and infestations) | 1 (1) | 0
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0
Pain - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) — BTX-A: Pain of skin; Skin pain. Placebo: Pain of skin; Stiff neck.
Pain::Back (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Pain::Head/headache (Nervous system disorders) | 1 (1) | 0
Pain::Pain NOS (General disorders) | 1 (1) | 1 (1) — BTX-A: Skin pain. Placebo: Pain of skin r/t biopsy
Vomiting (Gastrointestinal disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No